CLINICAL TRIAL: NCT06042322
Title: Retrospective Analysis of Pain in Patients Who Receive a Nerve Block for Surgery
Brief Title: Retrospective Analysis of Pain After Nerve Block in Surgical Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Yun-Yun K. Chen, Principal Investigator, Brigham and Women's Hospital
Other Study IDs: 2023P000514
Record Dates: First submitted 2023-08-29; First posted 2023-09-18 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Regional Anesthesia Morbidity; Acute Pain; Knee Osteoarthritis
MeSH Terms: conditions — Acute Pain; Osteoarthritis, Knee | interventions — Early Intervention, Educational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TKA with nerve block no intervention: Patients who received a single shot adductor canal nerve block prior to total knee arthroplasty surgery January 2017-June 2018
- TKA with nerve block with intervention: Patients who received a single shot adductor canal nerve block prior to total knee arthroplasty surgery during March 2019-March 2020, and received an educational intervention
  Interventions: Other: Educational intervention

INTERVENTIONS:
Other: Educational intervention — Multidisciplinary educational intervention was performed by orthopedic, anesthesia, and nursing team. This included a discussion of the patient's pain plan and a patient visit.
  Groups: TKA with nerve block with intervention

SUMMARY:
This is a retrospective study looking at patients who received a nerve block for surgery and assessing pain after the nerve block resolves, with or without an educational intervention, over two periods of time.

DETAILED DESCRIPTION:
Regional anesthesia (RA) is a vital tool that can serve as the primary anesthetic or as part of a multimodal perioperative pain regimen. RA is strongly associated with decreased acute and persistent pain and opioid consumption postoperatively. However, some patients experience an acute worsening of pain into the severe range around the time of RA resolution, also known as "rebound pain" (RP). The incidence of RP has been reported as high as 40-50% after a single shot nerve block for patients undergoing ambulatory surgery.

This retrospective study aims to look at patients who received a nerve block for surgery and assessing pain after the nerve block resolves in the presence and absence of certain interventions, such as a multidisciplinary educational intervention.

The investigators will assess patients who received a primary total knee arthroplasty who received a single shot adductor canal nerve block, received pericapsular injection by the surgeon, and had a length of stay > 16 hours.

ELIGIBILITY:
Inclusion Criteria:

* primary total knee arthroplasty
* received an adductor canal nerve block
* received pericapsular injection by surgeon intraoperatively
* admitted for overnight stay and > 16 hours post-nerve block

Exclusion Criteria:

* age < 18
* prior total knee arthroplasty on ipsilateral knee

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Using the Mass General Brigham Enterprise Data Warehouse, electronic health record data will be retrieved: adult patients, 18 years of age or older, who received a primary total knee arthroplasty, an adductor canal nerve block, pericapsular injection, and admitted to stay overnight (>16 hours post nerve block).
Sampling Method: Non-Probability Sample
Enrollment: 166 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Difference in maximum pain score, 0-10; (0 = no pain, 10 = worst pain) | 6-24 hours
  Difference in maximum pain score, numerical pain rating scale 0-10, 6-24 hours after nerve block between the two cohorts

SECONDARY OUTCOMES:
Average pain score 0-10; (0 = no pain, 10 = worst pain) | 6-24 hours
  Difference in area under the curve of pain scores, numerical pain rating scale 0-10, 6-24 hours after nerve block between the two cohorts (educational intervention and non-educational intervention time periods)
Difference in incidence of rebound pain | 6-24 hours
  Difference in incidence pain score ≥ 7 between 6-24 hours post nerve block between the two cohorts
Comparison of evening opioids given | 6-24 hours
  Comparison of if evening opioids were or were not given (yes/no) between the two cohorts
Difference in total opioids given | 6-24 hours
  Difference in total opioids given (mEq of morphine) between the two cohorts
Difference in length of stay | 0-2 years
  Difference in length of stay (days) between the two cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Yun K Chen, MD, Principal Investigator — Brigham and Women's Hospital